CLINICAL TRIAL: NCT06501040
Title: Increasing Knowledge and Interest in Cancer Clinical Trials
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hayley Thompson (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Hayley Thompson, Hayley Thompson. Ph.D., Barbara Ann Karmanos Cancer Institute
Organization: Barbara Ann Karmanos Cancer Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2019-137; NCI-2020-07119 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-137 (Other: Wayne State University/Karmanos Cancer Institute); P30CA022453 (NIH)
Record Dates: First submitted 2024-05-03; First posted 2024-07-15 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Educational Status; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Health Services Research (educational video) (Experimental): Participants view educational video consisting of information on the purpose of clinical trials, myths associated with clinical trials, and how to find more information about clinical trials.
  Interventions: Other: Web-based Educational Intervention; Other: Questionnaire Administration

INTERVENTIONS:
Other: Web-based Educational Intervention — View web-based educational video
  Other Names: Education for Intervention
Other: Questionnaire Administration — Pre video baseline survey and a post video educational survey

SUMMARY:
This trial investigates how well a video-based clinical trial education session works in increasing knowledge and interest in cancer clinical trials among individuals in the metropolitan Detroit region of the Karmanos Cancer Institute (KCI) catchment area. This educational activity may help researchers learn more about individuals' awareness of clinical trials, knowledge, and intention to participates in a clinical trial.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To increase cancer clinical trial knowledge and interest through video-based education among individuals aged 21 and older in the metropolitan Detroit region of the KCI catchment area.

OUTLINE:

Participants view educational video consisting of information on the purpose of clinical trials, myths associated with clinical trials, and how to find more information about clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 21 and older
* Participants will be identified through Karmanos Cancer Institute's (KCI) clinical treatment center
* Participants will be identified through community-based KCI-sponsored events
* Participants will have voiced an interest to participate followed by an Informed consent

Exclusion Criteria

* none

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 384 (Estimated)
Dates: Start 2020-06-12 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Increase in Clinical Trial Awareness and Knowledge | Baseline and immediately post intervention up to 1 day
  An 11-question true and false questionnaire regarding Knowledge will be administered prior to and immediately after a video-based educational session on Clinical Trials

SECONDARY OUTCOMES:
Increase in intentions to participate in cancer clinical trials. | Baseline and immediately post intervention up to 1 day
  A 6-question standard Likert scale questionnaire regarding Intention will be administered prior to and immediately after a video-based educational session on Clinical Trials.

CONTACTS AND LOCATIONS:
Overall Officials: Hayley Thompson, Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Wayne State University/Karmanos Cancer Institute, Detroit, Michigan, United States